CLINICAL TRIAL: NCT00101777
Title: Ventilatory Physiology in Children at Risk for Anxiety
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020093; 02-M-0093
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Anxiety; Panic Disorder
Keywords: Anxiety; Ventilation; Panic Disorder; Children; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Respiratory Aspiration

SUMMARY:
The importance of the proposed research project derives from a steady accumulation of research findings on the relationship between respiration and anxiety. The relationship between panic disorder and abnormalities in respiration has been recognized for more than 10 years. Increased sensitivity to CO2 exposure in panic disorder represents the most consistent finding supporting this relationship. The current proposal follows naturally from three sets of recent research findings in the area of panic disorder. First, our group has recently shown that children with anxiety disorders, like adults with panic disorder, exhibit increased sensitivity to CO2. Second, other researchers have shown that psychiatrically healthy relatives of patients with panic disorder also exhibit increased sensitvity to CO2. Finally, our group has also recently shown that children of adults with panic disorder exhibit high rates of anxiety disorders, particularly separation anxiety disorder, the childhood anxiety disorder which exhibits the highest degree of CO2 sensitivity. These three findings suggest that children of parents with panic disorder may exhibit a latent vulnerability to panic disorder, manifested as increased sensitivity to CO2.

A secondary feature of the proposed research project derives from a steady accumulation of research findings in basic science literature outlining the parts of the brain that mediate fear and anxiety in animals. It may be possible to use insights from research on the brain basis of fear in animals to develop methods for assessing the brain basis of fear in humans. Moreover, work in animals notes changes in brain systems that mediate fear and anxiety across development. If development. If developmentally sensitive methods could be used to study fear in children, it may also be possible to greatly enhance our understanding of the manner in which the relationship between brain function and fear changes as children age. If similarities could be demonstrated across animals and humans in these areas, new insights on potential treatments for anxiety could be more readily transferred from the laboratory to the clinic. A second goal of the current proposal is to refine two neuropsychological probes that are thought to assess functional aspects of brain systems implicated in fear and anxiety across various species, from rodents to humans.

DETAILED DESCRIPTION:
The importance of the proposed research project derives from a steady accumulation of research findings on the relationship between respiration and anxiety. The relationship between panic disorder and abnormalities in respiration has been recognized for more than 10 years. Increased sensitivity to CO2 exposure in panic disorder represents the most consistent finding supporting this relationship. The current proposal follows naturally from three sets of recent research findings in the area of panic disorder. First, our group has recently shown that children with anxiety disorders, like adults with panic disorder, exhibit increased sensitivity to CO2. Second, other researchers have shown that psychiatrically healthy relatives of patients with panic disorder also exhibit increased sensitvity to CO2. Finally, our group has also recently shown that children of adults with panic disorder exhibit high rates of anxiety disorders, particularly separation anxiety disorder, the childhood anxiety disorder which exhibits the highest degree of CO2 sensitivity. These three findings suggest that children of parents with panic disorder may exhibit a latent vulnerability to panic disorder, manifested as increased sensitivity to CO2.

A secondary feature of the proposed research project derives from a steady accumulation of research findings in basic science literature outlining the parts of the brain that mediate fear and anxiety in animals. It may be possible to use insights from research on the brain basis of fear in animals to develop methods for assessing the brain basis of fear in humans. Moreover, work in animals notes changes in brain systems that mediate fear and anxiety across development. If developmentally sensitive methods could be used to study fear in children, it may also be possible to greatly enhance our understanding of the manner in which the relationship between brain function and fear changes as children age. If similarities could be demonstrated across animals and humans in these areas, new insights on potential treatments for anxiety could be more readily transferred from the laboratory to the clinic. A second goal of the current proposal is to refine two neuropsychological probes that are thought to assess functional aspects of brain systems implicated in fear and anxiety across various species, from rodents to humans.

ELIGIBILITY:
INCLUSION CRITERIA (ALL OFFSPRING):

Ages greater than or equal to 9 years 0 months.

Parent able to give written informed consent.

Offspring ages 12 years 0 months to 17 years 11 months able to give written assent.

Offspring ages 9 years 0 months to 11 years 11 months able to give verbal assent.

Offspring ages 18 years 0 months.

Absence of medical condition that will interfere with CO(2) procedure.

INCLUSION CRITERIA (PARENTS):

Has met DSM-IV criteria for one or more of the following disorders:

Panic Disorder

Social Phobia

Major Depressive Disorder

OR No Disorder.

EXCLUSION CRITERIA (ALL OFFSPRING):

Clinically significant or unstable medical disorders; cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine, hematological or other systemic disease.

History of mania, schizophrenia or other psychosis, or current serious suicidal ideation.

Females who are pregnant.

Children currently on medications that affect breathing.

IQ less than 70.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 479
Dates: Start 2001-12; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Papp LA, Klein DF, Martinez J, Schneier F, Cole R, Liebowitz MR, Hollander E, Fyer AJ, Jordan F, Gorman JM. Diagnostic and substance specificity of carbon-dioxide-induced panic. Am J Psychiatry. 1993 Feb;150(2):250-7. doi: 10.1176/ajp.150.2.250. PMID 8123056
- [Background] Papp LA, Martinez JM, Klein DF, Coplan JD, Norman RG, Cole R, de Jesus MJ, Ross D, Goetz R, Gorman JM. Respiratory psychophysiology of panic disorder: three respiratory challenges in 98 subjects. Am J Psychiatry. 1997 Nov;154(11):1557-65. doi: 10.1176/ajp.154.11.1557. PMID 9356564
- [Background] Perna G, Gabriele A, Caldirola D, Bellodi L. Hypersensitivity to inhalation of carbon dioxide and panic attacks. Psychiatry Res. 1995 Aug 28;57(3):267-73. doi: 10.1016/0165-1781(95)02723-a. PMID 7501737